CLINICAL TRIAL: NCT01196988
Title: Immunogenicity and Safety Study of GSK Biologicals' Influenza Vaccine GSK2321138A When Administered in Children
Brief Title: Immunogenicity and Safety Study of GSK Biologicals' Influenza Vaccine When Administered in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 113275
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2017-03

CONDITIONS: Influenza
Keywords: GSK Biologicals influenza vaccine GSK2321138A; influenza infection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- GSK2321138A 1 Group (Experimental): Subjects aged 3-17 years received if primed, 1 dose of GSK2321138A at Day 0 and if unprimed, 2 doses of GSK2321138A at Day 0 and Day 28. The vaccine was administered intramuscularly into the deltoid for subjects aged 12 months or above or into the anterolateral region of the thigh for subjects below 12 month of age. The vaccine was administered in the non-dominant side of the body at Day 0 and in the opposite side at Day 28.
  Interventions: Biological: Influenza vaccine GSK2321138A
- Fluarix Group (Active Comparator): Subjects aged 3-17 years received if primed, 1 dose of Fluarix at Day 0 and if unprimed, 2 doses of Fluarix at Day 0 and Day 28. The vaccine was administered intramuscularly into the deltoid for subjects aged 12 months or above or into the anterolateral region of the thigh for subjects below 12 month of age. The vaccine was administered in the non-dominant side of the body at Day 0 and in the opposite side at Day 28.
  Interventions: Biological: FluarixTM
- GSK2604409A Group (Active Comparator): Subjects aged 3-17 years received if primed, 1 dose of GSK2604409A at Day 0 and if unprimed, 2 doses of GSK2604409A at Day 0 and Day 28. The vaccine was administered intramuscularly into the deltoid for subjects aged 12 months or above or into the anterolateral region of the thigh for subjects below 12 month of age. The vaccine was administered in the non-dominant side of the body at Day 0 and in the opposite side at Day 28.
  Interventions: Biological: Influenza vaccine GSK2604409A
- GSK2321138A 2 Group (Experimental): Subjects aged 6-35 months received if primed, 1 dose of GSK2321138A at Day 0 and if unprimed, 2 doses of GSK2321138A at Day 0 and Day 28. The vaccine was administered intramuscularly into the deltoid for subjects aged 12 months or above or into the anterolateral region of the thigh for subjects below 12 month of age. The vaccine was administered in the non-dominant side of the body at Day 0 and in the opposite side at Day 28.
  Interventions: Biological: Influenza vaccine GSK2321138A

INTERVENTIONS:
Biological: Influenza vaccine GSK2321138A — intramuscular injections
  Arms: GSK2321138A 1 Group; GSK2321138A 2 Group
Biological: FluarixTM — intramuscular injections
  Arms: Fluarix Group
Biological: Influenza vaccine GSK2604409A — intramuscular injections
  Arms: GSK2604409A Group

SUMMARY:
This study is designed to assess the safety and immunogenicity of GlaxoSmithKline (GSK) Biologicals' investigational vaccine GSK2321138A in children aged 3 to 17 years, and to describe safety and immunogenicity of the GSK Biologicals' investigational vaccine GSK2321138A in children aged 6 to 35 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* For non US countries:
* - Children, male or female, aged between 6 months and 17 years at the time of the first study vaccination.

For US :

* Children, male or female, aged between 3 and 17 years at the time of the first study vaccination
* Written informed consent obtained from the subject parent(s) or LAR(s) of the subject. Assent obtained from the subject when applicable.
* Subjects in stable health as determined by investigator's clinical examination and assessment of subjects' medical history.
* Written informed assent obtained from the subject if/as required by local regulations.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* - has practiced adequate contraception for 30 days prior to vaccination,
* - and has a negative urine pregnancy test on the day of vaccination,
* - and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period. Routine registered childhood vaccinations are permitted.
* Planned administration of any vaccine 30 days prior and 30 days after any study vaccine administration.
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* Prior receipt of any seasonal or pandemic influenza vaccine (registered or investigational) within 6 months preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to enrolment in this study or planned administration during the study period.
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study, or planned during the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* History of seizures or progressive neurological disease.
* History of Guillain-Barré syndrome within 6 weeks of receipt of prior inactivated influenza virus vaccine.
* Concurrently participating in another clinical study, at any time during the study period in which the subject has been or will be exposed to an investigational or a non-investigational product .
* History of hypersensitivity to a previous dose of influenza vaccine, history of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines
* Acute disease and/or fever at the time of enrolment
* Ongoing aspirin therapy
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study
* Child in Care.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3027 (Actual)
Dates: Start 2010-10-04; Primary Completion 2011-06-15 (Actual); Study Completion 2011-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (56):
- United States (13):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Elmira, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Angelo, Texas
- Czechia (10):
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Humpolec
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Kolín
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Odolena Voda
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Tábor
- France (9):
  - GSK Investigational Site, Aix-en-Provence
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, La Bouëxière
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Seysses
  - GSK Investigational Site, Tours
- Germany (22):
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Gilching, Bavaria
  - GSK Investigational Site, Kirchheim, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Weimar, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Philippines (2):
  - GSK Investigational Site, Dasmariñas, Cavite
  - GSK Investigational Site, Quezon City

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Domachowske JB, Pankow-Culot H, Bautista M, Feng Y, Claeys C, Peeters M, Innis BL, Jain V. A randomized trial of candidate inactivated quadrivalent influenza vaccine versus trivalent influenza vaccines in children aged 3-17 years. J Infect Dis. 2013 Jun 15;207(12):1878-87. doi: 10.1093/infdis/jit091. Epub 2013 Mar 7. PMID 23470848
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were differentiated according to their priming status. Primed subjects had received at least 1 dose of an influenza A (H1N1) 2009 monovalent vaccine and had received 2 doses of seasonal influenza in the last season or had received at least 1 dose prior to last season. Unprimed subjects had not.
Pre-assignment Details: 3015 subjects out of the 3027 who were enrolled in the study were vaccinated. Remaining subjects were not included in the participant flow as started as they failed to meet protocol criteria. The treatment was stratified by age strata: 3-8 and 9-17 years. Another arm evaluates the GSK2321138A vaccine for children aged 6-17 and 18-35 months.
Period: Overall Study
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Started | 915 | 912 | 911 | 277
Completed | 891 | 880 | 886 | 276
Not Completed | 24 | 32 | 25 | 1
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 4 | 0
Not completed — Lost to Follow-up | 16 | 29 | 21 | 1
Not completed — Other | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group | Total
Number analyzed (Participants) | 915 | 912 | 911 | 277 | 3015
Age, Continuous [Mean (Standard Deviation); unit: Months] | 98.5 (44.40) | 98.2 (45.50) | 99.6 (44.20) | 22.1 (8.02) | 79.6 (35.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 443 | 439 | 440 | 118 | 1440
  Male | 472 | 473 | 471 | 159 | 1575

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata).
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity which included all vaccinated and eligible subjects for whom data concerning Immunogenicity outcomes variables were available and for whom assay results were available for antibodies against at least one study vaccine component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 791 | 819 | 801 | 234
titers
  FLU A/Cal/7/09, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU A/Cal/7/09, PRE | 21.6 [19.7 to 23.7] | 24.9 [22.8 to 27.3] | 22.1 [20.1 to 24.2] | 12.3 [10.2 to 14.8]
  FLU A/Cal/7/09, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU A/Cal/7/09, POST | 386.2 [357.3 to 417.4] | 433.2 [401.0 to 468.0] | 422.3 [390.5 to 456.5] | 140.0 [113.7 to 172.3]
  FLU A/Vic/210/09, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU A/Vic/210/09, PRE | 29.0 [26.6 to 31.6] | 31.4 [28.8 to 34.2] | 31.2 [28.6 to 34.2] | 8.6 [7.4 to 9.9]
  FLU A/Vic/210/09, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU A/Vic/210/09, POST | 228.8 [215.0 to 243.4] | 227.3 [213.3 to 242.3] | 234.0 [219.1 to 249.9] | 87.5 [73.8 to 103.7]
  FLU B/Bri/60/08, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU B/Bri/60/08, PRE | 30.9 [28.2 to 33.9] | 31.0 [28.2 to 34.0] | 33.2 [30.2 to 36.6] | 9.0 [7.9 to 10.4]
  FLU B/Bri/60/08, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU B/Bri/60/08, POST | 244.2 [227.5 to 262.1] | 245.6 [229.2 to 263.2] | 88.4 [81.5 to 95.8] | 86.4 [72.6 to 102.9]
  FLU B/Bri/3/07, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU B/Bri/3/07, PRE | 77.3 [70.0 to 85.3] | 77.2 [70.0 to 85.2] | 84.7 [76.6 to 93.6] | 13.1 [11.4 to 15.2]
  FLU B/Bri/3/07, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU B/Bri/3/07, POST | 569.6 [533.6 to 608.1] | 224.7 [207.9 to 242.9] | 643.3 [603.2 to 686.1] | 167.7 [144.1 to 195.3]

2. Primary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata).
Time Frame: At Day 28 (for primed subjects) and Day 56 (for unprimed subjects)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 790 | 818 | 800 | 232
Participants
  FLU A/California/7/09 | 722 | 735 | 733 | 181
  FLU A/Victoria/210/09 | 571 | 578 | 575 | 159
  FLU B/Brisbane/60/08 | 553 | 560 | 237 | 158
  FLU B/Brisbane/3/07 | 573 | 303 | 566 | 191

3. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease by Age Strata.
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata).
  Subjects were assessed according to 2 age strata: 3-8 years and 9-17 years.
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 791 | 819 | 801
titers
  FLU A/Cal/7/09, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU A/Cal/7/09, PRE, 3-8 years | 20.7 [18.3 to 23.3] | 22.2 [19.8 to 24.9] | 22.4 [19.8 to 25.3]
  FLU A/Cal/7/09, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU A/Cal/7/09, POST, 3-8 years | 353.4 [319.9 to 390.3] | 382.1 [345.4 to 422.7] | 381.3 [345.0 to 421.5]
  FLU A/Cal/7/09, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Cal/7/09, PRE, 9-17 years | 23.2 [20.2 to 26.6] | 30.2 [26.1 to 34.9] | 21.5 [18.6 to 24.8]
  FLU A/Cal/7/09, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Cal/7/09, POST, 9-17 years | 445.8 [393.9 to 504.7] | 533.3 [474.9 to 599.0] | 502.0 [444.1 to 567.5]
  FLU A/Vic/210/09, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU A/Vic/210/09, PRE, 3-8 years | 29.3 [26.1 to 32.9] | 32.9 [29.2 to 37.0] | 31.5 [28.0 to 35.5]
  FLU A/Vic/210/09, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU A/Vic/210/09, POST, 3-8 years | 245.5 [226.4 to 266.2] | 242.0 [222.9 to 262.8] | 244.4 [224.1 to 266.5]
  FLU A/Vic/210/09, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Vic/210/09, PRE, 9-17 years | 28.5 [25.1 to 32.3] | 29.0 [25.8 to 32.7] | 30.8 [27.0 to 35.1]
  FLU A/Vic/210/09, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Vic/210/09, POST, 9-17 years | 204.1 [185.5 to 224.5] | 204.9 [185.4 to 226.6] | 217.5 [196.9 to 240.2]
  FLU B/Bri/60/08, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU B/Bri/60/08, PRE, 3-8 years | 27.1 [24.0 to 30.6] | 25.1 [22.3 to 28.3] | 27.9 [24.6 to 31.6]
  FLU B/Bri/60/08, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU B/Bri/60/08, POST, 3-8 years | 236.3 [215.4 to 259.2] | 222.3 [202.8 to 243.7] | 79.2 [71.2 to 88.2]
  FLU B/Bri/60/08, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/60/08, PRE, 9-17 years | 38.3 [33.4 to 43.9] | 43.9 [38.2 to 50.6] | 44.7 [38.6 to 51.7]
  FLU B/Bri/60/08, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/60/08, POST, 9-17 years | 257.5 [230.7 to 287.5] | 289.8 [262.1 to 320.4] | 106.4 [94.6 to 119.8]
  FLU B/Bri/3/07, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU B/Bri/3/07, PRE, 3-8 years | 54.9 [48.7 to 61.9] | 51.9 [45.9 to 58.7] | 57.6 [50.9 to 65.1]
  FLU B/Bri/3/07, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU B/Bri/3/07, POST, 3-8 years | 481.3 [443.2 to 522.8] | 163.5 [148.4 to 180.1] | 566.7 [522.9 to 614.1]
  FLU B/Bri/3/07, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/3/07, PRE, 9-17 years | 134.3 [115.2 to 156.5] | 149.3 [130.3 to 171.1] | 162.8 [140.4 to 188.6]
  FLU B/Bri/3/07, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/3/07, POST, 9-17 years | 748.1 [676.9 to 826.8] | 380.6 [342.1 to 423.4] | 797.9 [719.5 to 885.0]

4. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease by Age Strata.
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata).
  Subjects were assessed according to 2 age strata: 6-17 months and 18-35 months.
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK2321138A 2 Group
Number analyzed (Participants) | 234
titers
  FLU A/Cal/7/09, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU A/Cal/7/09, PRE, 6-17 months | 7.1 [5.5 to 9.1]
  FLU A/Cal/7/09, POST, 6-17 months: number analyzed (Participants) | 71
  FLU A/Cal/7/09, POST, 6-17 months | 56.2 [39.9 to 79.2]
  FLU A/Cal/7/09, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU A/Cal/7/09, PRE, 18-35 months | 15.6 [12.3 to 19.8]
  FLU A/Cal/7/09, POST, 18-35 months: number analyzed (Participants) | 163
  FLU A/Cal/7/09, POST, 18-35 months | 208.3 [164.6 to 263.4]
  FLU A/Vic/210/09, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU A/Vic/210/09, PRE, 6-17 months | 6.2 [5.1 to 7.6]
  FLU A/Vic/210/09, POST, 6-17 months: number analyzed (Participants) | 71
  FLU A/Vic/210/09, POST, 6-17 months | 43.8 [33.7 to 57.0]
  FLU A/Vic/210/09, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU A/Vic/210/09, PRE, 18-35 months | 9.8 [8.1 to 11.9]
  FLU A/Vic/210/09, POST, 18-35 months: number analyzed (Participants) | 163
  FLU A/Vic/210/09, POST, 18-35 months | 118.2 [96.8 to 144.4]
  FLU B/Bri/60/08, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU B/Bri/60/08, PRE, 6-17 months | 5.9 [5.3 to 6.6]
  FLU B/Bri/60/08, POST, 6-17 months: number analyzed (Participants) | 71
  FLU B/Bri/60/08, POST, 6-17 months | 40.2 [31.2 to 51.6]
  FLU B/Bri/60/08, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU B/Bri/60/08, PRE, 18-35 months | 10.8 [9.0 to 13.1]
  FLU B/Bri/60/08, POST, 18-35 months: number analyzed (Participants) | 163
  FLU B/Bri/60/08, POST, 18-35 months | 120.7 [98.2 to 148.4]
  FLU B/Bri/3/07, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU B/Bri/3/07, PRE, 6-17 months | 10.0 [7.9 to 12.7]
  FLU B/Bri/3/07, POST, 6-17 months: number analyzed (Participants) | 71
  FLU B/Bri/3/07, POST, 6-17 months | 93.5 [73.5 to 119.0]
  FLU B/Bri/3/07, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU B/Bri/3/07, PRE, 18-35 months | 14.8 [12.4 to 17.7]
  FLU B/Bri/3/07, POST, 18-35 months: number analyzed (Participants) | 163
  FLU B/Bri/3/07, POST, 18-35 months | 216.3 [180.9 to 258.7]

5. Secondary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza Disease by Age Strata.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata). Subjects were assessed according to 2 age strata: 3-8 years and 9-17 years.
Time Frame: At Day 28 (for primed subjects) and Day 56 (for unprimed subjects)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 790 | 818 | 800
Participants
  FLU A/California/7/09, 3-8 years: number analyzed (Participants) | 488 | 510 | 503
  FLU A/California/7/09, 3-8 years | 447 | 468 | 457
  FLU A/California/7/09, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/California/7/09, 9-17 years | 275 | 267 | 276
  FLU A/Victoria/210/09, 3-8 years: number analyzed (Participants) | 488 | 510 | 503
  FLU A/Victoria/210/09, 3-8 years | 367 | 365 | 376
  FLU A/Victoria/210/09, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Victoria/210/09, 9-17 years | 204 | 213 | 199
  FLU B/Brisbane/60/08, 3-8 years: number analyzed (Participants) | 488 | 510 | 503
  FLU B/Brisbane/60/08, 3-8 years | 364 | 367 | 154
  FLU B/Brisbane/60/08, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Brisbane/60/08, 9-17 years | 189 | 193 | 83
  FLU B/Brisbane/3/07, 3-8 years: number analyzed (Participants) | 488 | 510 | 503
  FLU B/Brisbane/3/07, 3-8 years | 376 | 203 | 403
  FLU B/Brisbane/3/07, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Brisbane/3/07, 9-17 years | 197 | 100 | 163

6. Secondary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza Disease by Age Strata.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata). Subjects were assessed according to 2 age strata: 6-17 months and 18-35 months.
Time Frame: At Day 28 (for primed subjects) and Day 56 (for unprimed subjects)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 2 Group
Number analyzed (Participants) | 232
Participants
  FLU A/California/7/09, 6-17 months: number analyzed (Participants) | 70
  FLU A/California/7/09, 6-17 months | 43
  FLU A/California/7/09, 18-35 months: number analyzed (Participants) | 162
  FLU A/California/7/09, 18-35 months | 138
  FLU A/Victoria/210/09, 6-17 months: number analyzed (Participants) | 70
  FLU A/Victoria/210/09, 6-17 months | 37
  FLU A/Victoria/210/09, 18-35 months: number analyzed (Participants) | 162
  FLU A/Victoria/210/09, 18-35 months | 122
  FLU B/Brisbane/60/08, 6-17 months: number analyzed (Participants) | 70
  FLU B/Brisbane/60/08, 6-17 months | 36
  FLU B/Brisbane/60/08, 18-35 months: number analyzed (Participants) | 162
  FLU B/Brisbane/60/08, 18-35 months | 122
  FLU B/Brisbane/3/07, 6-17 months: number analyzed (Participants) | 70
  FLU B/Brisbane/3/07, 6-17 months | 52
  FLU B/Brisbane/3/07, 18-35 months: number analyzed (Participants) | 162
  FLU B/Brisbane/3/07, 18-35 months | 139

7. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata).
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 791 | 819 | 801 | 234
Participants
  FLU A/California/7/09, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU A/California/7/09, PRE | 343 | 404 | 353 | 60
  FLU A/California/7/09, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU A/California/7/09, POST | 764 | 793 | 778 | 187
  FLU A/Victoria/210/09, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU A/Victoria/210/09, PRE | 381 | 412 | 409 | 34
  FLU A/Victoria/210/09, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU A/Victoria/210/09, POST | 775 | 800 | 773 | 169
  FLU B/Brisbane/60/08, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU B/Brisbane/60/08, PRE | 381 | 396 | 399 | 28
  FLU B/Brisbane/60/08, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU B/Brisbane/60/08, POST | 770 | 790 | 639 | 167
  FLU B/Brisbane/3/07, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU B/Brisbane/3/07, PRE | 565 | 575 | 593 | 48
  FLU B/Brisbane/3/07, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU B/Brisbane/3/07, POST | 785 | 772 | 798 | 212

8. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease by Age Strata.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata). Subjects were assessed according to 2 age strata: 3-8 years and 9-17 years.
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 791 | 819 | 801
Participants
  FLU A/Cal/7/09, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU A/Cal/7/09, PRE, 3-8 years | 206 | 234 | 230
  FLU A/Cal/7/09, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU A/Cal/7/09, POST, 3-8 years | 469 | 491 | 487
  FLU A/Cal/7/09, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Cal/7/09, PRE, 9-17 years | 137 | 170 | 123
  FLU A/Cal/7/09, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Cal/7/09, POST, 9-17 years | 295 | 302 | 291
  FLU A/Vic/210/09, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU A/Vic/210/09, PRE, 3-8 years | 253 | 277 | 269
  FLU A/Vic/210/09, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU A/Vic/210/09, POST, 3-8 years | 477 | 496 | 481
  FLU A/Vic/210/09, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Vic/210/09, PRE, 9-17 years | 128 | 135 | 140
  FLU A/Vic/210/09, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Vic/210/09, POST, 9-17 years | 298 | 304 | 292
  FLU B/Bri/60/08, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU B/Bri/60/08, PRE, 3-8 years | 217 | 218 | 232
  FLU B/Bri/60/08, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU B/Bri/60/08, POST, 3-8 years | 478 | 489 | 378
  FLU B/Bri/60/08, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/60/08, PRE, 9-17 years | 164 | 178 | 167
  FLU B/Bri/60/08, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/60/08, POST, 9-17 years | 292 | 301 | 261
  FLU B/Bri/3/07, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU B/Bri/3/07, PRE, 3-8 years | 315 | 309 | 329
  FLU B/Bri/3/07, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU B/Bri/3/07, POST, 3-8 years | 485 | 465 | 503
  FLU B/Bri/3/07, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/3/07, PRE, 9-17 years | 250 | 266 | 264
  FLU B/Bri/3/07, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/3/07, POST, 9-17 years | 300 | 307 | 295

9. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease by Age Strata.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata). Subjects were assessed according to 2 age strata: 6-17 months and 18-35 months.
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 2 Group
Number analyzed (Participants) | 234
Participants
  FLU A/Cal/7/09, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU A/Cal/7/09, PRE, 6-17 months | 6
  FLU A/Cal/7/09, POST, 6-17 months: number analyzed (Participants) | 71
  FLU A/Cal/7/09, POST, 6-17 months | 45
  FLU A/Cal/7/09, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU A/Cal/7/09, PRE, 18-35 months | 54
  FLU A/Cal/7/09, POST, 18-35 months: number analyzed (Participants) | 163
  FLU A/Cal/7/09, POST, 18-35 months | 142
  FLU A/Vic/210/09, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU A/Vic/210/09, PRE, 6-17 months | 4
  FLU A/Vic/210/09, POST, 6-17 months: number analyzed (Participants) | 71
  FLU A/Vic/210/09, POST, 6-17 months | 39
  FLU A/Vic/210/09, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU A/Vic/210/09, PRE, 18-35 months | 30
  FLU A/Vic/210/09, POST, 18-35 months: number analyzed (Participants) | 163
  FLU A/Vic/210/09, POST, 18-35 months | 130
  FLU B/Bri/60/08, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU B/Bri/60/08, PRE, 6-17 months | 1
  FLU B/Bri/60/08, POST, 6-17 months: number analyzed (Participants) | 71
  FLU B/Bri/60/08, POST, 6-17 months | 38
  FLU B/Bri/60/08, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU B/Bri/60/08, PRE, 18-35 months | 27
  FLU B/Bri/60/08, POST, 18-35 months: number analyzed (Participants) | 163
  FLU B/Bri/60/08, POST, 18-35 months | 129
  FLU B/Bri/3/07, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU B/Bri/3/07, PRE, 6-17 months | 11
  FLU B/Bri/3/07, POST, 6-17 months: number analyzed (Participants) | 71
  FLU B/Bri/3/07, POST, 6-17 months | 61
  FLU B/Bri/3/07, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU B/Bri/3/07, PRE, 18-35 months | 37
  FLU B/Bri/3/07, POST, 18-35 months: number analyzed (Participants) | 163
  FLU B/Bri/3/07, POST, 18-35 months | 151

10. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:80. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata).
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 791 | 819 | 801 | 234
Participants
  FLU A/California/7/09, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU A/California/7/09, PRE | 201 | 218 | 202 | 49
  FLU A/California/7/09, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU A/California/7/09, POST | 732 | 763 | 744 | 155
  FLU A/Victoria/210/09, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU A/Victoria/210/09, PRE | 228 | 245 | 267 | 27
  FLU A/Victoria/210/09, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU A/Victoria/210/09, POST | 721 | 748 | 721 | 125
  FLU B/Brisbane/60/08, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU B/Brisbane/60/08, PRE | 244 | 258 | 269 | 18
  FLU B/Brisbane/60/08, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU B/Brisbane/60/08, POST | 708 | 733 | 488 | 140
  FLU B/Brisbane/3/07, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU B/Brisbane/3/07, PRE | 454 | 462 | 476 | 24
  FLU B/Brisbane/3/07, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU B/Brisbane/3/07, POST | 779 | 692 | 784 | 175

11. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease by Age Strata.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:80. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata). Subjects were assessed according to 2 age strata: 3-8 years and 9-17 years.
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 791 | 819 | 801
Participants
  FLU A/Cal/7/09, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU A/Cal/7/09, PRE, 3-8 years | 130 | 128 | 141
  FLU A/Cal/7/09, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU A/Cal/7/09, POST, 3-8 years | 453 | 471 | 464
  FLU A/Cal/7/09, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Cal/7/09, PRE, 9-17 years | 71 | 90 | 61
  FLU A/Cal/7/09, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Cal/7/09, POST, 9-17 years | 279 | 292 | 280
  FLU A/Vic/210/09, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU A/Vic/210/09, PRE, 3-8 years | 156 | 177 | 190
  FLU A/Vic/210/09, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU A/Vic/210/09, POST, 3-8 years | 446 | 462 | 446
  FLU A/Vic/210/09, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Vic/210/09, PRE, 9-17 years | 72 | 68 | 77
  FLU A/Vic/210/09, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Vic/210/09, POST, 9-17 years | 275 | 286 | 275
  FLU B/Bri/60/08, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU B/Bri/60/08, PRE, 3-8 years | 145 | 140 | 150
  FLU B/Bri/60/08, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU B/Bri/60/08, POST, 3-8 years | 430 | 441 | 286
  FLU B/Bri/60/08, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/60/08, PRE, 9-17 years | 99 | 118 | 119
  FLU B/Bri/60/08, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/60/08, POST, 9-17 years | 278 | 292 | 202
  FLU B/Bri/3/07, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU B/Bri/3/07, PRE, 3-8 years | 233 | 227 | 248
  FLU B/Bri/3/07, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU B/Bri/3/07, POST, 3-8 years | 480 | 395 | 493
  FLU B/Bri/3/07, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/3/07, PRE, 9-17 years | 221 | 235 | 228
  FLU B/Bri/3/07, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/3/07, POST, 9-17 years | 299 | 297 | 291

12. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease by Age Strata.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:80. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata). Subjects were assessed according to 2 age strata: 6-17 months and 18-35 months.
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 2 Group
Number analyzed (Participants) | 234
Participants
  FLU A/California/7/09, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU A/California/7/09, PRE, 6-17 months | 6
  FLU A/California/7/09, POST, 6-17 months: number analyzed (Participants) | 71
  FLU A/California/7/09, POST, 6-17 months | 31
  FLU A/California/7/09, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU A/California/7/09, PRE, 18-35 months | 43
  FLU A/California/7/09, POST, 18-35 months: number analyzed (Participants) | 163
  FLU A/California/7/09, POST, 18-35 months | 124
  FLU A/Victoria/210/09, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU A/Victoria/210/09, PRE, 6-17 months | 4
  FLU A/Victoria/210/09, POST, 6-17 months: number analyzed (Participants) | 71
  FLU A/Victoria/210/09, POST, 6-17 months | 18
  FLU A/Victoria/210/09, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU A/Victoria/210/09, PRE, 18-35 months | 23
  FLU A/Victoria/210/09, POST, 18-35 months: number analyzed (Participants) | 163
  FLU A/Victoria/210/09, POST, 18-35 months | 107
  FLU B/Brisbane/60/08, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU B/Brisbane/60/08, PRE, 6-17 months | 0
  FLU B/Brisbane/60/08, POST, 6-17 months: number analyzed (Participants) | 71
  FLU B/Brisbane/60/08, POST, 6-17 months | 25
  FLU B/Brisbane/60/08, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU B/Brisbane/60/08, PRE, 18-35 months | 18
  FLU B/Brisbane/60/08, POST, 18-35 months: number analyzed (Participants) | 163
  FLU B/Brisbane/60/08, POST, 18-35 months | 115
  FLU B/Brisbane/3/07, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU B/Brisbane/3/07, PRE, 6-17 months | 4
  FLU B/Brisbane/3/07, POST, 6-17 months: number analyzed (Participants) | 71
  FLU B/Brisbane/3/07, POST, 6-17 months | 43
  FLU B/Brisbane/3/07, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU B/Brisbane/3/07, PRE, 18-35 months | 20
  FLU B/Brisbane/3/07, POST, 18-35 months: number analyzed (Participants) | 163
  FLU B/Brisbane/3/07, POST, 18-35 months | 132

13. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:120. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata).
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 791 | 819 | 801 | 234
Participants
  FLU A/California/7/09, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU A/California/7/09, PRE | 71 | 92 | 79 | 28
  FLU A/California/7/09, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU A/California/7/09, POST | 669 | 720 | 690 | 122
  FLU A/Victoria/210/09, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU A/Victoria/210/09, PRE | 103 | 124 | 121 | 15
  FLU A/Victoria/210/09, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU A/Victoria/210/09, POST | 597 | 597 | 599 | 82
  FLU B/Brisbane/60/08, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU B/Brisbane/60/08, PRE | 123 | 126 | 148 | 9
  FLU B/Brisbane/60/08, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU B/Brisbane/60/08, POST | 578 | 607 | 300 | 83
  FLU B/Brisbane/3/07, PRE: number analyzed (Participants) | 790 | 819 | 800 | 232
  FLU B/Brisbane/3/07, PRE | 300 | 324 | 327 | 7
  FLU B/Brisbane/3/07, POST: number analyzed (Participants) | 791 | 818 | 801 | 234
  FLU B/Brisbane/3/07, POST | 730 | 564 | 756 | 129

14. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease by Age Strata.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:120. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata). Subjects were assessed according to 2 age strata: 3-8 years and 9-17 years.
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 791 | 819 | 801
Participants
  FLU A/Cal/7/09, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU A/Cal/7/09, PRE, 3-8 years | 47 | 56 | 57
  FLU A/Cal/7/09, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU A/Cal/7/09, POST, 3-8 years | 410 | 442 | 428
  FLU A/Cal/7/09, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Cal/7/09, PRE, 9-17 years | 24 | 36 | 22
  FLU A/Cal/7/09, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Cal/7/09, POST, 9-17 years | 259 | 278 | 262
  FLU A/Vic/210/09, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU A/Vic/210/09, PRE, 3-8 years | 70 | 92 | 87
  FLU A/Vic/210/09, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU A/Vic/210/09, POST, 3-8 years | 380 | 385 | 390
  FLU A/Vic/210/09, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Vic/210/09, PRE, 9-17 years | 33 | 32 | 34
  FLU A/Vic/210/09, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Vic/210/09, POST, 9-17 years | 217 | 212 | 209
  FLU B/Bri/60/08, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU B/Bri/60/08, PRE, 3-8 years | 75 | 66 | 82
  FLU B/Bri/60/08, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU B/Bri/60/08, POST, 3-8 years | 349 | 357 | 174
  FLU B/Bri/60/08, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/60/08, PRE, 9-17 years | 48 | 60 | 66
  FLU B/Bri/60/08, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/60/08, POST, 9-17 years | 229 | 250 | 126
  FLU B/Bri/3/07, PRE, 3-8 years: number analyzed (Participants) | 488 | 511 | 503
  FLU B/Bri/3/07, PRE, 3-8 years | 135 | 155 | 150
  FLU B/Bri/3/07, POST, 3-8 years: number analyzed (Participants) | 489 | 510 | 504
  FLU B/Bri/3/07, POST, 3-8 years | 444 | 301 | 473
  FLU B/Bri/3/07, PRE, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/3/07, PRE, 9-17 years | 165 | 169 | 177
  FLU B/Bri/3/07, POST, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Bri/3/07, POST, 9-17 years | 286 | 263 | 283

15. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease by Age Strata.
Description: A seroprotected subject was defined as as a vaccinated subject who had a serum HI titer ≥ 1:120. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata). Subjects were assessed according to 2 age strata: 6 -17 months and 18-35 months.
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 2 Group
Number analyzed (Participants) | 234
Participants
  FLU A/California/7/09, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU A/California/7/09, PRE, 6-17 months | 5
  FLU A/California/7/09, POST, 6-17 months: number analyzed (Participants) | 71
  FLU A/California/7/09, POST, 6-17 months | 18
  FLU A/California/7/09, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU A/California/7/09, PRE, 18-35 months | 23
  FLU A/California/7/09, POST, 18-35 months: number analyzed (Participants) | 163
  FLU A/California/7/09, POST, 18-35 months | 104
  FLU A/Victoria/210/09, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU A/Victoria/210/09, PRE, 6-17 months | 3
  FLU A/Victoria/210/09, POST, 6-17 months: number analyzed (Participants) | 71
  FLU A/Victoria/210/09, POST, 6-17 months | 11
  FLU A/Victoria/210/09, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU A/Victoria/210/09, PRE, 18-35 months | 12
  FLU A/Victoria/210/09, POST, 18-35 months: number analyzed (Participants) | 163
  FLU A/Victoria/210/09, POST, 18-35 months | 71
  FLU B/Brisbane/60/08, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU B/Brisbane/60/08, PRE, 6-17 months | 0
  FLU B/Brisbane/60/08, POST, 6-17 months: number analyzed (Participants) | 71
  FLU B/Brisbane/60/08, POST, 6-17 months | 7
  FLU B/Brisbane/60/08, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU B/Brisbane/60/08, PRE, 18-35 months | 9
  FLU B/Brisbane/60/08, POST, 18-35 months: number analyzed (Participants) | 163
  FLU B/Brisbane/60/08, POST, 18-35 months | 76
  FLU B/Brisbane/3/07, PRE, 6-17 months: number analyzed (Participants) | 70
  FLU B/Brisbane/3/07, PRE, 6-17 months | 1
  FLU B/Brisbane/3/07, POST, 6-17 months: number analyzed (Participants) | 71
  FLU B/Brisbane/3/07, POST, 6-17 months | 25
  FLU B/Brisbane/3/07, PRE, 18-35 months: number analyzed (Participants) | 162
  FLU B/Brisbane/3/07, PRE, 18-35 months | 6
  FLU B/Brisbane/3/07, POST, 18-35 months: number analyzed (Participants) | 163
  FLU B/Brisbane/3/07, POST, 18-35 months | 104

16. Secondary Outcome: Mean Geometric Increase (MGI) Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease.
Description: MGI is defined as the geometric mean of the within subject ratios of the post-vaccination reciprocal HI titer to the Day 0 reciprocal HI titer. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata).
Time Frame: At Day 28 (for primed subjects) and Day 56 (for unprimed subjects)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 790 | 818 | 800 | 232
fold change
  FLU A/California/7/09 | 18.0 [16.6 to 19.5] | 17.4 [16.0 to 18.8] | 19.2 [17.7 to 20.9] | 11.7 [10.2 to 13.4]
  FLU A/Victoria/210/09 | 7.9 [7.3 to 8.6] | 7.2 [6.7 to 7.8] | 7.5 [6.9 to 8.1] | 10.4 [9.0 to 11.9]
  FLU B/Brisbane/60/08 | 7.9 [7.3 to 8.6] | 7.9 [7.2 to 8.6] | 2.7 [2.5 to 2.9] | 9.7 [8.5 to 11.2]
  FLU B/Brisbane/3/07 | 7.4 [6.8 to 8.0] | 2.9 [2.7 to 3.1] | 7.6 [7.0 to 8.3] | 12.9 [11.0 to 15.3]

17. Secondary Outcome: Mean Geometric Increase (MGI) Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease by Age Strata.
Description: MGI is defined as the geometric mean of the within subject ratios of the post-vaccination reciprocal HI titer to the Day 0 reciprocal HI titer. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata). Subjects were assessed according to 2 age strata: 3-8 years and 9-17 years.
Time Frame: At Day 28 (for primed subjects) and Day 56 (for unprimed subjects)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 790 | 818 | 800
fold change
  FLU A/California/7/09, 3-8 years: number analyzed (Participants) | 488 | 510 | 503
  FLU A/California/7/09, 3-8 years | 17.2 [15.6 to 19.0] | 17.2 [15.6 to 18.9] | 17.2 [15.6 to 18.9]
  FLU A/California/7/09, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/California/7/09, 9-17 years | 19.2 [16.7 to 22.2] | 17.7 [15.2 to 20.5] | 23.3 [20.3 to 26.9]
  FLU A/Victoria/210/09, 3-8 years: number analyzed (Participants) | 488 | 510 | 503
  FLU A/Victoria/210/09, 3-8 years | 8.4 [7.6 to 9.3] | 7.3 [6.6 to 8.1] | 7.8 [7.1 to 8.5]
  FLU A/Victoria/210/09, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU A/Victoria/210/09, 9-17 years | 7.2 [6.2 to 8.2] | 7.1 [6.2 to 8.1] | 7.1 [6.2 to 8.1]
  FLU B/Brisbane/60/08, 3-8 years: number analyzed (Participants) | 488 | 510 | 503
  FLU B/Brisbane/60/08, 3-8 years | 8.8 [7.9 to 9.8] | 8.8 [7.9 to 9.8] | 2.8 [2.6 to 3.1]
  FLU B/Brisbane/60/08, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Brisbane/60/08, 9-17 years | 6.7 [5.8 to 7.8] | 6.6 [5.7 to 7.6] | 2.4 [2.1 to 2.7]
  FLU B/Brisbane/3/07, 3-8 years: number analyzed (Participants) | 488 | 510 | 503
  FLU B/Brisbane/3/07, 3-8 years | 8.8 [7.9 to 9.8] | 3.1 [2.9 to 3.4] | 9.9 [8.9 to 11.0]
  FLU B/Brisbane/3/07, 9-17 years: number analyzed (Participants) | 302 | 308 | 297
  FLU B/Brisbane/3/07, 9-17 years | 5.6 [4.9 to 6.3] | 2.5 [2.3 to 2.8] | 4.9 [4.3 to 5.6]

18. Secondary Outcome: Mean Geometric Increase (MGI) Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease by Age Strata.
Description: MGI is defined as the geometric mean of the within subject ratios of the post-vaccination reciprocal HI titer to the Day 0 reciprocal HI titer. The 4 influenza strains assessed were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (Victoria) and FLU B/Brisbane/3/07 (Yamagata). Subjects were assessed according to 2 age strata: 6 -17 months and 18-35 months.
Time Frame: At Day 28 (for primed subjects) and Day 56 (for unprimed subjects)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | GSK2321138A 2 Group
Number analyzed (Participants) | 232
fold change
  FLU A/California/7/09, 6-17 months: number analyzed (Participants) | 70
  FLU A/California/7/09, 6-17 months | 8.2 [6.4 to 10.6]
  FLU A/California/7/09, 18-35 months: number analyzed (Participants) | 162
  FLU A/California/7/09, 18-35 months | 13.7 [11.7 to 16.0]
  FLU A/Victoria/210/09, 6-17 months: number analyzed (Participants) | 70
  FLU A/Victoria/210/09, 6-17 months | 7.3 [5.9 to 9.0]
  FLU A/Victoria/210/09, 18-35 months: number analyzed (Participants) | 162
  FLU A/Victoria/210/09, 18-35 months | 12.1 [10.2 to 14.3]
  FLU B/Brisbane/60/08, 6-17 months: number analyzed (Participants) | 70
  FLU B/Brisbane/60/08, 6-17 months | 6.9 [5.4 to 8.9]
  FLU B/Brisbane/60/08, 18-35 months: number analyzed (Participants) | 162
  FLU B/Brisbane/60/08, 18-35 months | 11.3 [9.6 to 13.2]
  FLU B/Brisbane/3/07, 6-17 months: number analyzed (Participants) | 70
  FLU B/Brisbane/3/07, 6-17 months | 9.5 [7.0 to 12.8]
  FLU B/Brisbane/3/07, 18-35 months: number analyzed (Participants) | 162
  FLU B/Brisbane/3/07, 18-35 months | 14.8 [12.2 to 18.0]

19. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling at the injection site. Any = incidence of a particular symptom regardless of intensity grade. Grade 3 pain = Cried when limb was moved/spontaneously painful (Child <6 years) or pain that prevented normal activity (Child >6 years). Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of the injection site.
Time Frame: During the 7-day (Days 0-6) follow-up period after any vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, on vaccinated subjects with available results and with the symptom completed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 903 | 902 | 906 | 277
Participants
  Any Pain | 444 | 425 | 416 | 116
  Grade 3 Pain | 20 | 21 | 13 | 5
  Any Redness | 225 | 214 | 206 | 100
  Grade 3 Redness | 12 | 3 | 6 | 1
  Any Swelling | 196 | 193 | 160 | 67
  Grade 3 Swelling | 11 | 10 | 3 | 0

20. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms in Subjects Younger Than 6 Years Old.
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and temperature [axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of any solicited general symptom regardless of intensity grade or relation to vaccination. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 irritability = crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite = not eating at all. Related = general symptom assessed by the investigator as causally related to the study vaccination. Grade 3 temperature = temperature >39.0°C.
Time Frame: During the 7-day (Days 0-6) follow-up period after any vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, on vaccinated subjects with available results and with the symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 291 | 314 | 280 | 277
Participants
  Any Drowsiness | 67 | 55 | 59 | 84
  Grade 3 Drowsiness | 5 | 3 | 2 | 7
  Related Drowsiness | 44 | 31 | 36 | 57
  Any Irritability | 65 | 56 | 53 | 119
  Grade 3 Irritability | 4 | 2 | 3 | 11
  Related Irritability | 44 | 37 | 31 | 81
  Any Loss of appetite | 59 | 40 | 47 | 83
  Grade 3 Loss of appetite | 3 | 3 | 3 | 12
  Related Loss of appetite | 37 | 24 | 25 | 50
  Temperature ≥37.5°C | 50 | 51 | 41 | 81
  Temperature >39°C | 4 | 2 | 3 | 18
  Related Temperature | 24 | 29 | 16 | 37

21. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms in Subjects Aged 6 Years or Older.
Description: as for outcome 20
Time Frame: During the 7-day (Days 0-6) follow-up period after any vaccination.
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group
Number analyzed (Participants) | 613 | 589 | 626
Participants
  Any Fatigue | 129 | 118 | 114
  Grade 3 Fatigue | 9 | 8 | 4
  Related Fatigue | 95 | 81 | 76
  Any Gastro. | 66 | 62 | 52
  Grade 3 Gastro. | 7 | 4 | 2
  Related Gastro. | 31 | 29 | 26
  Any Headache | 110 | 125 | 114
  Grade 3 Headache | 8 | 4 | 5
  Related Headache | 66 | 75 | 71
  Any Joint Pain | 69 | 63 | 51
  Grade 3 Joint Pain | 2 | 4 | 2
  Related Joint Pain | 44 | 43 | 36
  Any Muscle aches | 116 | 106 | 106
  Grade 3 Muscle aches | 4 | 8 | 3
  Related Muscle aches | 84 | 81 | 87
  Any Shivering | 44 | 31 | 37
  Grade 3 Shivering | 3 | 3 | 1
  Related Shivering | 27 | 23 | 22
  Temperature ≥37.5°C | 48 | 60 | 47
  Temperature >39°C | 7 | 5 | 3
  Related Temperature | 25 | 30 | 32

22. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3 = unsolicited AE that prevented normal activity Related = unsolicited AE assessed by the investigator as related to the vaccination.
Time Frame: During the 28-day (Days 0-27) follow-up period after any vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, on vaccinated subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 915 | 912 | 911 | 277
Participants
  Subjects with any AE(s) | 284 | 305 | 308 | 167
  Subjects with grade 3 AE(s) | 20 | 37 | 26 | 20
  Subjects with related AE(s) | 18 | 19 | 23 | 5

23. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Medically Attended Adverse Events (MAEs).
Description: MAEs were defined as AEs that resulted in medical attention (defined as hospitalization, an emergency room visit or a visit to or from medical personnel for any reason). Any = any MAE regardless of intensity or relationship to vaccination. Grade 3 MAE = MAE which prevented normal, everyday activities. Related = MAE assessed by the investigator as related to the vaccination. Assessment of intensity for MAEs was not performed.
Time Frame: During the entire study period (Day 0 - Day 180)
Population: The analysis was performed on the Total Vaccinated cohort, on vaccinated subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 915 | 912 | 911 | 277
Participants
  Subjects with any MAE(s) | 271 | 278 | 303 | 171
  Subjects with related MAE(s) | 2 | 4 | 4 | 2
  Subjects with Grade 3 MAE(s) | NA — Analysis was not performed. | NA — Analysis was not performed. | NA — Analysis was not performed. | NA — Analysis was not performed.

24. Secondary Outcome: Number of Subjects With Any and Related Potential Immune-Mediated Diseases (pIMDs).
Description: pIMDs were defined as a subset of AEs that included both clearly autoimmune diseases (AID) and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology.
Time Frame: During the entire study period (Day 0 - Day 180)
Population: The analysis was performed on the Total Vaccinated cohort, on vaccinated subjects with available results
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 915 | 912 | 911 | 277
Participants
  Subjects with any pIMD(s) | 0 | 0 | 2 | 0
  Subjects with related pIMD(s) | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (Day 0 - Day 180)
Population: The analysis was performed on the Total Vaccinated cohort, on vaccinated subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 915 | 912 | 911 | 277
Participants
  Subjects with any SAE(s) | 8 | 6 | 7 | 9
  Subjects with related SAE(s) | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Days With Solicited Local Symptoms.
Description: The number of days with any grade of local symptoms after Dose 1 and Dose 2 vaccination respectively was tabulated. Assessed solicited local symptoms for duration were pain, redness and swelling at the injection site.
Time Frame: During the 7-day (Days 0-6) follow-up period after vaccination.
Population: as for outcome 20
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 395 | 382 | 365 | 94
days
  Pain, Dose 1 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Pain, Dose 2: number analyzed (Participants) | 175 | 156 | 160 | 70
  Pain, Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Redness, Dose 1: number analyzed (Participants) | 208 | 192 | 189 | 84
  Redness, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.5 to 4.0]
  Redness, Dose 2: number analyzed (Participants) | 75 | 80 | 76 | 69
  Redness, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Swelling, Dose 1: number analyzed (Participants) | 167 | 155 | 135 | 44
  Swelling, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Swelling, Dose 2: number analyzed (Participants) | 70 | 65 | 59 | 39
  Swelling, Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]

27. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any grade of local symptoms after Dose 1 and Dose 2 vaccination respectively was tabulated. Assessed solicited general symptoms for duration were drowsiness, fatigue, gastrointestinal symptoms (Gastro.), headache, irritability, loss of appetite, muscle aches, shivering and temperature [axillary temperature equal to or above 37.5 degrees Celsius (°C)].
Time Frame: During the 7-day (Days 0-6) follow-up period after vaccination.
Population: as for outcome 20
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Number analyzed (Participants) | 121 | 113 | 99 | 79
days
  Drowsiness, Dose 1: number analyzed (Participants) | 50 | 39 | 38 | 66
  Drowsiness, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Drowsiness, Dose 2: number analyzed (Participants) | 29 | 29 | 32 | 45
  Drowsiness, Dose 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Fatigue, Dose 1: number analyzed (Participants) | 121 | 109 | 99 | 79
  Fatigue, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — Symptom not assessed in this group.
  Fatigue, Dose 2: number analyzed (Participants) | 33 | 25 | 33 | 79
  Fatigue, Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Gastro., Dose 1: number analyzed (Participants) | 60 | 56 | 45 | 79
  Gastro., Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Gastro., Dose 2: number analyzed (Participants) | 11 | 9 | 8 | 79
  Gastro., Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Headache, Dose 1: number analyzed (Participants) | 100 | 113 | 95 | 79
  Headache, Dose 1 | 1.0 [1.0 to 2.5] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Headache, Dose 2: number analyzed (Participants) | 19 | 21 | 29 | 79
  Headache, Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Irritability, Dose 1: number analyzed (Participants) | 49 | 42 | 40 | 79
  Irritability, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Irritability, Dose 2: number analyzed (Participants) | 37 | 33 | 27 | 79
  Irritability, Dose 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Joint pain, Dose 1: number analyzed (Participants) | 60 | 55 | 46 | 79
  Joint pain, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Joint pain, Dose 2: number analyzed (Participants) | 18 | 14 | 10 | 79
  Joint pain, Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Loss of appetite, Dose 1: number analyzed (Participants) | 45 | 29 | 25 | 56
  Loss of appetite, Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0] | 3.0 [1.0 to 4.5]
  Loss of appetite, Dose 2: number analyzed (Participants) | 22 | 26 | 26 | 50
  Loss of appetite, Dose 2 | 3.0 [1.0 to 4.0] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 3.0 [2.0 to 4.0]
  Muscle aches, Dose 1: number analyzed (Participants) | 107 | 94 | 99 | 79
  Muscle aches, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Muscle aches, Dose 2: number analyzed (Participants) | 25 | 20 | 19 | 79
  Muscle aches, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Shivering, Dose 1: number analyzed (Participants) | 39 | 26 | 31 | 79
  Shivering, Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 5.0] | 1.0 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Shivering, Dose 2: number analyzed (Participants) | 7 | 6 | 7 | 79
  Shivering, Dose 2 | 1.0 [1.0 to 3.0] | 1.5 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | NA [NA to NA] — Symptom not assessed in this group.
  Temperature, Dose 1: number analyzed (Participants) | 63 | 78 | 61 | 45
  Temperature, Dose 1 | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Temperature, Dose 2: number analyzed (Participants) | 40 | 44 | 33 | 53
  Temperature, Dose 2 | 1.5 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]

ADVERSE EVENTS:
Time Frame: SAE(s): during the entire study period (Day 0 - Day 180); Solicited local and general symptoms: during the 7-day (Days 0-6) follow-up period after any vaccination, Unsolicited AE(s): during the 28-day follow-up period (Days 0 to 27) after any vaccination.
Description: No reported SAE was assessed as related to study vaccination. For systematically assessed other AEs, the number of participants at risk included those from Total Vaccinated cohort with symptom sheet completed.
Arm/Group | GSK2321138A 1 Group | Fluarix Group | GSK2604409A Group | GSK2321138A 2 Group
Serious Adverse Events (participants affected / at risk) | 8/915 | 6/912 | 7/911 | 9/277
Other Adverse Events (participants affected / at risk) | 630/915 | 616/912 | 620/911 | 237/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2321138A 1 Group (N=915) | Fluarix Group (N=912) | GSK2604409A Group (N=911) | GSK2321138A 2 Group (N=277)
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Amoebiasis (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 3
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 2
Dengue fever (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 2
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK2321138A 1 Group (N=915) | Fluarix Group (N=912) | GSK2604409A Group (N=911) | GSK2321138A 2 Group (N=277)
Nasopharyngitis (Infections and infestations) | 49 | 60 | 64 | 37
Upper respiratory tract infection (Infections and infestations) | 48 | 51 | 46 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 40 | 36 | 45 | 21
Pyrexia (General disorders) | 23 | 23 | 28 | 18
Bronchitis (Infections and infestations) | 13 | 5 | 12 | 29
Fatigue (General disorders) | 129/613 | 118/589 | 114/626 | 0 — This result is for subjects 6 years old or older
Gastrointestinal (General disorders) | 66/613 | 62/589 | 52/626 | 0 — This result is for subjects 6 years old or older
Headache (General disorders) | 110/613 | 125/589 | 114/626 | 0 — This result is for subjects 6 years old or older
Joint Pain (General disorders) | 69/613 | 63/589 | 51/626 | 0 — This result is for subjects 6 years old or older
Muscle aches (General disorders) | 116/613 | 106/589 | 106/626 | 0 — This result is for subjects 6 years old or older
Temperature (Axillary) (General disorders) | 48/613 | 60/589 | 47/626 | 0 — This result is for subjects 6 years old or older
Irritability (General disorders) | 65/291 | 56/314 | 53/280 | 119 — This result is for subjects younger than 6 years old
Drowsiness (General disorders) | 67/291 | 55/314 | 59/280 | 84 — This result is for subjects younger than 6 years old
Loss of appetite (General disorders) | 59/291 | 40/314 | 47/280 | 83 — This result is for subjects younger than 6 years old
Pain (General disorders) | 444/903 | 425/902 | 416/906 | 116
Redness (General disorders) | 225/903 | 214/902 | 206/906 | 100
Swelling (General disorders) | 196/903 | 193/902 | 160/906 | 67
Temperature (Axillary) (General disorders) | 50/291 | 51/314 | 41/280 | 81 — This result is for subjects younger than 6 years old
Shivering (General disorders) | 44/613 | 31/589 | 37/626 | 0 — This result is for subjects 6 years old or older

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.